CLINICAL TRIAL: NCT03376971
Title: Real-Time Optical Biopsy for Improved Lung Cancer Diagnosis
Brief Title: Real-Time Optical Biopsy in Improving Lung Cancer Diagnosis in Patients Undergoing Lung Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1706540415; 1706540415 (Other: The University of Arizona)
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Lesion; Lung Cancer; Diagnoses Disease
Keywords: Lesion; Lung; Cancer; Diagnosis; Optical Biopsy; Biopsy
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Disease | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (lung biopsy) (Experimental): Patients undergo extraction of up to 3 additional lung biopsies from target lesions that are at least 2-3 cm in diameter using the 19 gauge SuperCore biopsy needle or the 20 gauge Rotax needle. The extracted tissue is imaged via confocal fluorescence microscopy using a variety of fluorescent contrast agents, such as fluorescein sodium, methylene blue, indocyanine green and then undergo hematoxylin and eosin processing.
  Interventions: Procedure: Biopsy; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biopsy — Undergo lung biopsy
  Other Names: Bx
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot early phase I trial studies how well real-time optical biopsy works in improving lung cancer diagnosis in patients undergoing lung biopsy. Real-time optical biopsy using confocal microscopy may improve the ability of physicians to diagnose lung cancer and accurately differentiate cancerous and benign lesions found during computed tomography screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Show that it is possible to distinguish lung cancer from benign lesions in ex vivo tissue samples using optical microscopy.

II. Test a proof-of-concept endoscopic instrument for imaging through a biopsy needle under computed tomography (CT) guidance on ex vivo tissue samples.

OUTLINE:

Patients undergo extraction of up to 3 additional lung biopsies from target lesions that are at least 2-3 cm in diameter using the 19 gauge SuperCore biopsy needle or the 20 gauge Rotax needle. The extracted tissue is imaged via confocal fluorescence microscopy using a variety of fluorescent contrast agents, such as, fluorescein sodium, methylene blue, or indocyanine green and then undergo hematoxylin and eosin processing.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be drawn from the pool of patients who have suspicious lesions identified on CT and who are already scheduled for a lung biopsy procedure with Dr. Woodhead or one of his colleagues
* Patients will be asked to consent to 2 to 3 extra biopsy samples to be used for this research project

Exclusion Criteria:

- Excluded from this study will be minors below age 18, prisoners, pregnant women, patients with a contraindication for additional lung biopsies, and patients who cannot give informed consent (language barrier, cognitive impairment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Diagnosis of ex vivo tissue samples for lung cancer or benign lesions using optical microscopy | At the time of biopsy
  The aim is to show that it is possible to distinguish lung cancer from benign lesions in ex vivo tissue samples using optical microscopy.
Imaging of ex vivo tissue samples using an endoscopic instrument | At the time of biopsy
  A proof-of-concept endoscopic instrument will be tested for imaging through a biopsy needle under computed tomography guidance on ex vivo tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rouse, PhD, Principal Investigator — The University of Arizona; Gregory Woodhead, MD, Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided